CLINICAL TRIAL: NCT00138879
Title: Plasma Citrulline Level: A Simple, Sensitive Method to Assess and Monitor Small Bowel Absorptive Function in Patients With Crohn's Disease?
Brief Title: Citrulline: A Plasmatic Marker to Assess and Monitor Small Bowel Crohn's Disease Patients
Status: Completed | Type: Observational
Sponsor: St Mark's Hospital Foundation (Other)
Other Study IDs: EC3155
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-08

CONDITIONS: Crohn's Disease; Short Bowel Syndrome; Malabsorption Syndromes; Celiac Disease
Keywords: Citrulline; Parenteral Nutrition; functioning intestinal mass; small bowel permeability and absorption; Granulomatous Enteritis
MeSH Terms: conditions — Crohn Disease; Short Bowel Syndrome; Malabsorption Syndromes; Celiac Disease; Hyperphagia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Citrulline is an amino acid produced in the intestine and in the liver, but the liver does not contribute significantly to circulating citrulline concentrations. The intestine is thus the only organ that normally releases significant amounts of citrulline into the blood. The investigators have designed a study looking at the value of measuring plasma citrulline concentration in patients with Crohn's disease and short bowel or normal intestinal length. Measuring the plasma citrulline concentration in short bowel patients may help to distinguish between patients who need permanent parenteral feeding from patients with just transient intestinal dysfunction. It may also help the investigators in understanding the small bowel intestinal length remaining and the absorptive integrity. In patients with normal intestinal length and Crohn's disease, it may be a reliable marker of small bowel damage and could be applied to establish therapeutic improvements. It has been demonstrated to strongly correlate (inversely) with severity on intestinal biopsies.

The investigators hypothesise that the plasma citrulline concentration is a marker for small bowel absorptive integrity and an appropriate surrogate for functional length of the small intestine.

Controlled data do not yet exist to establish the place of plasma citrulline in the assessment of small bowel function in man.

DETAILED DESCRIPTION:
Preliminary studies reported that plasma citrulline concentrations may be a reliable biochemical marker for intestinal dysfunction and absorptive enterocyte mass. The relationship between citrulline concentration and intestinal function has been supported in other studies including those examining rejection in small bowel allografts. Concentrations of citrulline are dramatically reduced in cases of mucosal damage (e.g. moderate graft rejection or viral enteritis) and strongly correlate (inversely) with severity on biopsy. Plasma citrulline concentration is lower also in patients with villous atrophy (24±13 μmol/L) than in healthy subjects (40±10 μmol/L) and patients with anorexia nervosa (39±9).

A citrulline threshold of 20 µmol/L apparently permitted the classification of short bowel syndrome patients into either transient or permanent intestinal failure categories, with 92% sensitivity, 90% specificity, and 95% positive and 86% negative predictive values, respectively. Experimental studies have been carried out also in assessing the value of citrulline as a marker for severity of small bowel epithelial damage from radiation. The plasma citrulline was shown to be a simple, non-invasive and sensitive assay to monitor and quantify radiation-induced small bowel damage in mice and humans. Otherwise, the literature on citrulline as a potential marker of intestinal and nutritional integrity is young and data for specific conditions come only from single centres; there are limited data on normal ranges. More crucially, however, there has been no attempt to clarify the effect of inflammation on citrulline homeostasis. To date there is no information in respect of patients with intestinal failure in whom there has been no resection.

We hypothesise that plasma citrulline concentration reflects small bowel absorptive capacity and correlates to the functional intestinal length independently from inflammation.

Comparisons: To exclude the possibility that citrulline merely reflects inflammation, control groups (six subjects each) with short bowel syndrome without inflammation (mesenteric infarct) (negative control); and those with inflammation but no anatomical loss (active coeliac disease) (positive controls); will be studied as well as healthy volunteers.

The study is designed to utilise patients from the positive and negative control groups to permit a correlation of plasma citrulline with intestinal length and with a "gold standard" assessment of intestinal function as judged from the patients need for nutritional intervention (from normal diet to dependence on home parenteral nutrition).

Plasma citrulline will be determined by Reverse-phase High Performance Liquid Chromatography (RF-HPLC) after an overnight fast. Albumin and Routine biochemical assessment will also be performed. Gastrointestinal permeability will be determined from the double sugar test using rhamnose and lactulose, and functional absorptive capacity will be estimated by D-Xylose absorption rate.

Analysis will allow for paired comparison between patients and between groups. Differences in the clinical performance of the various parameters will be determined. The study has adequate statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease (CD) with massive small bowel resection at least 24 months previously (< 50cm remaining)
* Crohn's disease with small bowel resection at least 24 months previously (50-150cm remaining)
* CD with no resection
* Mesenteric infarction with massive resection > 24 months previously (< 50cm remaining)
* Mesenteric infarction with massive resection > 24 months previously (50-150cm remaining); coeliac disease.
* Healthy volunteers.
* Body mass index within the normal range

Exclusion Criteria:

* Patients with surgical resection of stomach, duodenum or pancreas; or upper gastrointestinal (UGI) bypass.
* Oral feeding > 1.0-fold the estimated basal metabolic rate as assessed using Harris and Benedict equations.
* Patients with fistulating Crohn's disease
* Patients on steroids
* Patients with other important disease, which may interfere with the study (especially diabetes and renal impairment). Alcoholism, drug abuse or any other circumstances, which may compromise the patient's ability to comply with the study requirements.
* Pregnancy.
* Corticosteroid use or octreotide during, or in, the month before the study.
* Use of glucagon-like peptide 2 (GLP2), growth hormone (GH) or glutamine or triglycerides.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2003-05; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, Medicine, Study Chair — University College, London; Roy A. Sherwood, Biochemistry, Study Director — King's College Hospital NHS Trust; Cinzia Papadia, Medicine, Principal Investigator — Imperial College University of London
Locations (1):
- St Mark's Hospital, London, Middlesex, United Kingdom

REFERENCES:
- [Background] Blijlevens NM, Lutgens LC, Schattenberg AV, Donnelly JP. Citrulline: a potentially simple quantitative marker of intestinal epithelial damage following myeloablative therapy. Bone Marrow Transplant. 2004 Aug;34(3):193-6. doi: 10.1038/sj.bmt.1704563. PMID 15170165
- [Background] Lutgens LC, Deutz NE, Gueulette J, Cleutjens JP, Berger MP, Wouters BG, von Meyenfeldt MF, Lambin P. Citrulline: a physiologic marker enabling quantitation and monitoring of epithelial radiation-induced small bowel damage. Int J Radiat Oncol Biol Phys. 2003 Nov 15;57(4):1067-74. doi: 10.1016/s0360-3016(03)00781-8. PMID 14575838
- [Background] Pappas PA, Tzakis AG, Saudubray JM, Gaynor JJ, Carreno MR, Huijing F, Kleiner G, Rabier D, Kato T, Levi DM, Nishida S, Gelman B, Thompson JF, Mittal N, Ruiz P. Trends in serum citrulline and acute rejection among recipients of small bowel transplants. Transplant Proc. 2004 Mar;36(2):345-7. doi: 10.1016/j.transproceed.2003.12.007. PMID 15050154
- [Background] Selvaggi G, Weppler D, Tzakis A. Liver and gastrointestinal transplantation at the University of Miami. Clin Transpl. 2003:255-66. PMID 15387117
- [Background] Pappas PA, G Tzakis A, Gaynor JJ, Carreno MR, Ruiz P, Huijing F, Kleiner G, Rabier D, Kato T, Levi DM, Nishida S, Gelman B, Thompson JF, Mittal N, Saudubray JM. An analysis of the association between serum citrulline and acute rejection among 26 recipients of intestinal transplant. Am J Transplant. 2004 Jul;4(7):1124-32. doi: 10.1111/j.1600-6143.2004.00469.x. PMID 15196071
- [Background] Pappas PA, Saudubray JM, Tzakis AG, Rabier D, Carreno MR, Gomez-Marin O, Huijing F, Gelman B, Levi DM, Nery JR, Kato T, Mittal N, Nishida S, Thompson JF, Ruiz P. Serum citrulline as a marker of acute cellular rejection for intestinal transplantation. Transplant Proc. 2002 May;34(3):915-7. doi: 10.1016/s0041-1345(02)02668-4. No abstract available. PMID 12034237
- [Background] Crenn P, Vahedi K, Lavergne-Slove A, Cynober L, Matuchansky C, Messing B. Plasma citrulline: A marker of enterocyte mass in villous atrophy-associated small bowel disease. Gastroenterology. 2003 May;124(5):1210-9. doi: 10.1016/s0016-5085(03)00170-7. PMID 12730862
- [Background] Crenn P, Coudray-Lucas C, Thuillier F, Cynober L, Messing B. Postabsorptive plasma citrulline concentration is a marker of absorptive enterocyte mass and intestinal failure in humans. Gastroenterology. 2000 Dec;119(6):1496-505. doi: 10.1053/gast.2000.20227. PMID 11113071
- [Background] Windmueller HG, Spaeth AE. Source and fate of circulating citrulline. Am J Physiol. 1981 Dec;241(6):E473-80. doi: 10.1152/ajpendo.1981.241.6.E473. PMID 7325229
- [Background] Nightingale JM, Bartram CI, Lennard-Jones JE. Length of residual small bowel after partial resection: correlation between radiographic and surgical measurements. Gastrointest Radiol. 1991 Fall;16(4):305-6. doi: 10.1007/BF01887374. PMID 1936771
- [Background] D'Antiga L, Dhawan A, Davenport M, Mieli-Vergani G, Bjarnason I. Intestinal absorption and permeability in paediatric short-bowel syndrome: a pilot study. J Pediatr Gastroenterol Nutr. 1999 Nov;29(5):588-93. doi: 10.1097/00005176-199911000-00021. PMID 10554128
- [Background] Detsky AS, McLaughlin JR, Baker JP, Johnston N, Whittaker S, Mendelson RA, Jeejeebhoy KN. What is subjective global assessment of nutritional status? JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):8-13. doi: 10.1177/014860718701100108. PMID 3820522
- [Background] Zhang WZ, Kaye DM. Simultaneous determination of arginine and seven metabolites in plasma by reversed-phase liquid chromatography with a time-controlled ortho-phthaldialdehyde precolumn derivatization. Anal Biochem. 2004 Mar 1;326(1):87-92. doi: 10.1016/j.ab.2003.11.006. PMID 14769339
- [Background] Sherwood RA. Amino acid measurement by high-performance liquid chromatography using electrochemical detection. J Neurosci Methods. 1990 Sep;34(1-3):17-22. doi: 10.1016/0165-0270(90)90037-g. PMID 2259239
- [Background] Sherwood RA, Titheradge AC, Richards DA. Measurement of plasma and urine amino acids by high-performance liquid chromatography with electrochemical detection using phenylisothiocyanate derivatization. J Chromatogr. 1990 Jun 29;528(2):293-303. doi: 10.1016/s0378-4347(00)82388-9. PMID 2384569